CLINICAL TRIAL: NCT06020872
Title: My Meal Plate - Promoting the Health Literacy of Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: En-Chi Chiu (Other)
Collaborators: Taiwan Adventist Hospital (Other)
Responsible Party: Sponsor-Investigator, En-Chi Chiu, Associate Professor, National Taipei University of Nursing and Health Sciences
Organization: National Taipei University of Nursing and Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 109-E-20
Record Dates: First submitted 2023-08-24; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Nutrition, Healthy
Keywords: health literacy

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health literacy group (Experimental): Participants received the health literacy related to healthy plate.
  Interventions: Other: Health literacy program
- Control group (No Intervention): Participants did not receive the health literacy related to healthy plate.

INTERVENTIONS:
Other: Health literacy program — Health literacy program was the health education related to healthy plate.
  Arms: Health literacy group

SUMMARY:
This study was to investigate the results on health literacy through the program of my meal plate.

DETAILED DESCRIPTION:
Subjects were randomized to the intervention group and control group. The primary outcome was the Health Literacy on my Plate.

ELIGIBILITY:
Inclusion Criteria:

* patients who have ordered the general diet of the hospital and took more than three meals in a row.

Exclusion Criteria:

* pregnant woman
* unconscious
* people who cannot read

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Health Eating Literacy questionnaire | 30 minutes
  The Health Eating Literacy questionnaire is to assess person's ability to understand and remember on the healthcare information related to healthy eating principles.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Chi Lin, MS, Principal Investigator — Taiwan Adventist Hospital
Locations (1):
- Taiwan Adventist Hospital, Taipei, Songshan District, Taiwan

IPD SHARING:
Plan to Share IPD: No